CLINICAL TRIAL: NCT03346213
Title: Cardiopulmonary Exercise Testing Before and After Intravenous Iron: a Prospective Clinical Study
Brief Title: CArdio PulmOnary Exercise Testing and IntRAvenous Iron- 'CAPOEIRA-I STUDY'
Acronym: CAPOEIRA-I
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University College, London (Other); University of Bayreuth (Other)
Responsible Party: Sponsor
Other Study IDs: CRI
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Anemia; Anemia, Iron Deficiency
Keywords: Cardiopulmonary exercise testing; Intravenous iron; Total haemoglobin mass
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma stored in freezers at University Hospital Southampton
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major surgery: 1. Adult patients undergoing elective surgery
  2. Having a CPET as part of routine care
  3. Patients with a Hb value of < 130 g/L who are iron deficient, iron restricted/deplete or have functional iron deficiency.
  4. Able to provide written informed consent.
  Interventions: Drug: MonoFer

INTERVENTIONS:
Drug: MonoFer — Anaemic patients undergoing major surgery who would routinely be receiving intravenous iron 'MonoFer' will get this as part of routine care. They will then have a CPET repeated at least 10 days afterwards.

SUMMARY:
Red blood cells contain a chemical called haemoglobin which carries oxygen from the lungs around the body. When the amount of haemoglobin is reduced, a patient is 'anaemic'. Anaemia can have many causes, but affects about a third of patients having major surgery in hospital. After their operation these anaemic patients are more likely to suffer serious complications. This may be because the body needs extra oxygen - and so enough haemoglobin - to heal and recover successfully from the trauma of surgery.

For a similar reason, patients' overall fitness before surgery is very important. Less fit patients are much more likely to get complications after surgery. To help us assess the risk of complications, the investigators measure patients' fitness before surgery using a cycling exercise test. The investigators monitor a number of things that show us how well the heart, the lungs and the muscles respond when they are under stress. People who are very anaemic tend to perform less well on this cycling test.

Anaemia is often due to a lack of iron, which helps make haemoglobin. Usually people get iron from foods such as red meat and spinach. Some conditions mean that patients lose iron, such as a tumour bleeding. Other illnesses make it difficult for the body to absorb iron from the gut in the first place. Both lead to a state of low iron in the body and eventually this leads to anaemia. One way to treat anaemia quickly before surgery is to give iron into the bloodstream (intra-venous). It is thought that this might reduce the risk of complications after surgery, but it is not known whether this is because it improves overall fitness, or for other reasons.

The investigators plan to carry out a study called CAPOEIRA-I (CArdio PulmOnary Exercise testing and IntRAvenous Iron) to find out whether giving patients intravenous iron improves their fitness. The investigators will measure this by doing a cycle exercise test before and then at least 10 days after the iron is given. The investigators will also measure how much the total amount of haemoglobin chnages with iron treatment. Intravenous iron is already routinely used for these patients, so the only additional activity for the study is the extra exercise test, some extra blood tests and the measurement of haemoglobin after the iron has taken effect.

DETAILED DESCRIPTION:
Anaemia is common in the elective surgical population, a prevalence of around 30% being consistently reported in large cohorts.

Cardiopulmonary exercise testing (CPET), which provides an objective assessment of aerobic fitness by measuring oxygen consumption (O2) and carbon dioxide production is widely considered the gold standard assessment of functional capacity as it dynamically tests the pulmonary, cardiovascular and musculoskeletal system and their interplay in a single test. CPET parameters are affected by a number of patient factors including effort, ability to turn the pedals on an exercise bike, pulmonary function, and crucially oxygen delivery to the respiring tissues, which is dependent on blood oxygen content and flow to the tissues via cardiac output.

The oxygen carrying capacity of arterial blood is largely influenced by the haemoglobin content (or total haemoglobin mass (tHb-mass)). tHb-mass affects CPET performance to a greater degree than haemoglobin concentration ([Hb]). [Hb] is dependent on plasma volume (PV) and shows a greater fluctuation day to day than tHb-mass.

Studies in athletes show the detrimental affect of blood volume loss (i.e. deliberate venesection) and haemoglobin content loss on CPET performance. The corollary of this is illegal blood manipulation, which improves CPET performance. The same is seen post altitude training camps with increased tHb-mass leading to improved maximal exercise performance.

Aerobic capacity is defined as the maximum amount of oxygen that can be consumed by the body per unit time and is the gold standard measure of physical fitness. VO2max is classically defined as 'a plateau in oxygen uptake attained during maximal exercise despite further increases in exercise workload, thereby defining the limits of the cardiorespiratory system'. However, many individuals do not reach a plateau in oxygen uptake despite maximum exertion, and the term VO2peak is used instead. This is the highest measured oxygen consumption during exercise and is typically averaged over a 30 second period. O2 at anaerobic threshold (VO2AT) is defined as: 'the highest sustained intensity of exercise for which the measurement of oxygen uptake can account for the entire energy requirement.' An alternative definition is 'the exercise intensity at which lactate starts to accumulate in the blood stream above rest'. These oxygen uptake variables are in part dependent on the oxygen carrying capacity of the blood, which is in turn dependent on blood haemoglobin levels.

Major surgery places an increased metabolic demand on the body. Perhaps for this reason, both lower preoperative VO2peak and VO2AT values are associated with increased morbidity and mortality after major surgery. Much of the literature in this area is derived from studies reporting CPET variables. Given that the oxygen uptake variables VO2peak and VO2AT are positively correlated with tHb-mass, it may be that some of the physical fitness-outcome relationship is mediated through haemoglobin-related effects rather than cardiorespiratory function, providing a mechanistic basis to poor CPET performance in many patients with anaemia.

Few studies have examined the impact of blood manipulation - either transfusion or iron therapy - on CPET variables in patients. A study by Wright et al examined 20 patients with chronic anaemia due to 'stable haematological conditions' requiring blood transfusions. A CPET was performed before the blood transfusion and repeated 2-6 days after the transfusion of 1-4 units of blood (median 3). A mean rise in [Hb] from 8.3-11.2 g dl-1 was associated with a mean (SD) rise in O2AT from 10.4 (2.4) to 11.6 (2.5) mlkg-1min -1, (p= 0.018). (10). When corrected for the change in Hb concentration, the anaerobic threshold increased by a mean (SD) of 0.39 (0.74) ml kg-1 min-1 per g dl-1 Hb.

The results were consistent with a study in patients with beta thalassaemia major that compared exercise performance before, and 2 hours after haemotransfusion. Exercise duration increased from 7.3 (+/- 2.8) to 10.3 (+/- 2.3) minutes (p<0.05), and O2 peak increased from 28.5 (+/- 5.0) to 36.2 (+/- 7.1) ml kg-1min-1; (p<0.05).

Measuring haemoglobin concentration vs. total haemoglobin mass

Traditionally, the concentration of circulating haemoglobin [Hb] has been used as a clinical measure of the blood's oxygen carrying capacity. However, a low [Hb] may be due to a reduced amount of haemoglobin (absolute mass of circulating haemoglobin; tHb-mass) or an increased volume of dilution (plasma volume). Thus, [Hb] may be stable and tHb-mass low in the context of acute bleeding, [Hb] normal or elevated but tHb-mass low in the context of dehydration, or [Hb] low but tHb-mass normal or high in the context of excess plasma volume (fluid). Therefore, the use of [Hb] to define blood oxygen carrying capacity may be misleading under some circumstances.

tHb-mass represents the absolute mass of circulating haemoglobin in the body, the measured [Hb] being dependent upon tHb-mass and blood volume (BV) (sum of plasma volume (PV) and total red cell volume]). The proportion of oxygen carried in solution in plasma is trivial (0.3 ml per 100 ml of plasma) under normal physiological conditions, whereas each gram of Hb binds up to 1.39 mL of oxygen. Thus, tHb-mass is the principal determinant of total blood O2-carrying capacity and may provide additional information regarding the clinical status of patients than that provided by [Hb] alone.

Alternatively, a recently developed blood test capable of estimating absolute vascular volumes may be applied as a direct test to correct for any plasma volume fluctuations influencing a [Hb] value. As the model requires only a simple blood sample it may be a suitable alternative to estimate vascular volumes (and tHb-mass) if the patient is unable to perform the oCOR technique.

Classification of anaemia

The terminology around the classification of anaemia can be complex. There is no single laboratory parameter comprehensively reflecting the overall iron status of an individual. The POAS pathway used at UHS simplifies this (Appendix 1). In the perioperative period there are a number of possible causes of iron-related anaemia:

* Iron deficiency: Ferritin <30 g,l-1
* Iron deficiency and functional iron deficiency (FID) (ferritin 30-100g.l-1 with TSAT <20% and a CRP >5.
* Iron restriction/deplete Ferritin 30-100 with TSAT >20% or CRP raised/normal.
* If Ferritin is >100g,l-1 cause of anaemia could be non iron deficient anaemia or FID
* Functional iron deficiency: insufficient iron incorporation into erythroid precursors despite apparently adequate body iron stores. Recognised by the presence of stainable iron in the bone marrow, with a normal serum ferritin value,
* Anaemia of chronic inflammation: functional iron deficiency caused by chronic inflammation.
* A blood film is useful to detect iron deficiency alongside FID to determine which patients may benefit from iron therapy.

The investigators have defined how anaemia is classified and who would be eligible for intravenous iron therapy based on international consensus and local hospital guidelines. Patients who do not fall into the clear groups of iron deficiency, iron repletion or functional iron deficiency as per the POAS guidance are not suitable for intravenous iron and will not be eligible for this study.

Research statement

Preoperative anaemia is common, and is associated with poorer outcomes after major surgery. Impaired physical performance, as assessed by CPET, is likewise associated with impaired outcomes, and may be partly due to pre-operative anaemia.

The investigators wish to test the feasibility of performing a CPET test then administering intravenous iron and repeating a CPET prior to surgery in patients being considered for elective surgery. The investigators want to find out if treating anaemic patients who are suitable for intravenous iron therapy affects their CPET variables. This will help to inform further work to see if intravenous iron therapy combined with CPET adjusted risk stratification improves morbidity and/or mortality for anaemic patients undergoing major elective surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients undergoing elective surgery
2. Having a CPET as part of routine care
3. Patients with a Hb value of < 130 g/L who are iron deficient, iron restricted/deplete or have functional iron deficiency as described in 5.2 and Appendix 1
4. Able to provide written informed consent.

Patients with mixed aetiology anaemia who are either iron deficient, iron replete or functionally iron deficient alongside B12 or folate deficiency will be eligible for the study alongside treatment of their other nutritional deficiency.

Exclusion Criteria:

1. Pregnant women
2. Prisoners
3. Hypersensitivity to the active substance, to 'Monofer' (iron isomaltoside 1000) or any of its excipients
4. Known documented serious hypersensitivity to any parenteral iron products
5. Haemochromatosis or other iron overload states
6. Acute liver or renal failure
7. Active infection
8. Those receiving a blood transfusion between the CPET tests
9. Unable/ contraindication to perform CPET (Appendix 3)
10. Haemoglobinopathies such as Sickle Cell Anaemia or Thalassemia
11. Other cause for anaemia such as haematological malignancy, haemolysis, hypothyroidism.

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This cohort is composed of patients attending University Hospital Southampton NHS Foundation trust for major surgery who are found to be anaemic as part of routine clinical screening and are deemed suitable for intravenous iron therapy by the clinical team.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in oxygen consumption at anaerobic threshold (VO2AT) measured in mls/kg/min | Up to 6 weeks
  Using cardiopulmonary exercise testing (CPET) to assess the oxygen consumption at anaerobic threshold before and then after intravenous iron therapy.

SECONDARY OUTCOMES:
Change from baseline in peak oxygen consumption (VO2peak) measured in mls/kg/min | Up to 6 weeks
  Using cardiopulmonary exercise testing (CPET) to assess the oxygen consumption at peak exercise before and then after intravenous iron therapy therapy
Change from baseline haemoglobin concentration [Hb] measured in grams per litre (g.l-1) | Up to 6 weeks
  Laboratory measured haemoglobin concentration
Change from baseline in total haemoglobin mass measured in grams | Up to 6 weeks
  By using the optimised carbon monoxide rebreathing technique (oCOR) total haemoglobin mass will be measured before intravenous iron therapy and then again after intravenous iron therapy
Change form baseline in hepcidin assay measured in nanograms per millilitre (ng/ml) | Up to 6 weeks
  Hepcidin is iron regulatory hormone produced in the liver that affects iron transport. This will be measured twice.
Change form baseline in serum ferritin measured in micrograms per litre | Up to 6 weeks
  Ferritin is an acute phase protein but it is also the body major storage protein for iron.
Change form baseline in transferrin saturation (TSAT) (percentage) | Up to 6 weeks
  Plasma marker of iron storage and availability.
Change form baseline in serum iron measured in micromols per litre | Up to 6 weeks
  Plasma measure of iron availability.
Length of hospital stay in days | Up to 6 weeks
  Hospital length of stay after to include entire perioperative stay. (This is routinely collected already as part of the preoperative optimisation of anaemia before surgery (POAS) service.)

OTHER OUTCOMES:
Change from baseline- Creatinine | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Calcium | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Platelet count | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Low density lipoprotein | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Total protein | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Albumin | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Cholesterol | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Triglyceride | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Thyroxine | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Plateletcrit | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Neutrophils | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- White blood cell count | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.
Change from baseline- Monocytes | Up to 6 weeks
  Additional blood tests taken as part of the volume descriptive biomarker panel.

CONTACTS AND LOCATIONS:
Overall Officials: James Plumb, BMBS, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton NHS Foundation trust, Southampton, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside of the study team